CLINICAL TRIAL: NCT01238705
Title: Effect of Combined Antihypertensive Therapy on Blood Pressure and Sexual Function in Patients With Essential Hypertension
Brief Title: Combined Antihypertensive Therapy and Sexual Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LanZhou University (Other)
Responsible Party: Jing Yu, The Second Hospital of LanZhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0709TCYA068
Record Dates: First submitted 2010-10-12; First posted 2010-11-11 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Hypertension; Sexual Dysfunction
Keywords: Hypertension; Antihypertensive Agents; Combination; Sexual Dysfunction; Oxidative Stress
MeSH Terms: conditions — Hypertension; Sexual Dysfunction, Physiological | interventions — Felodipine; Irbesartan; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Felodipine,Irbesartan,Sexual Dysfunction (Active Comparator)
  Interventions: Drug: Felodipine add Irbesartan
- Felodipine,Metoprolol,Sexual Dysfunction (Active Comparator)
  Interventions: Drug: Felodipine add Metoprolol

INTERVENTIONS:
Drug: Felodipine add Irbesartan — Felodipine Sustained Release Tablets,5mg/day,AstraZeneca Pharmaceutical Co.Ltd., Registration Number: H20030415.
  Irbesartan,150mg/day, Sanofi - Aventis Pharmaceutical company, Registration Number: H20080074.
  Other Names: Plendil; Aprovel
  Arms: Felodipine,Irbesartan,Sexual Dysfunction
Drug: Felodipine add Metoprolol — Felodipine Sustained Release Tablets,5mg/day,AstraZeneca Pharmaceutical Co.Ltd., Registration Number: H20030415.
  Metoprolol Succinate,47.5mg/day,AstraZeneca Pharmaceutical Co.Ltd., Registration Number: J20050061.
  Other Names: Plendil; Betaloc
  Arms: Felodipine,Metoprolol,Sexual Dysfunction

SUMMARY:
This randomized,active controlled study aimed to compare the effects on sexual function of treatment with combined antihypertensive drugs.

The researchers hypothesize that:

1. Both felodipine-irbesartan combination and felodipine-metoprolol combination are effective in lowing blood pressure in patients with essential hypertension.
2. Felodipine-metoprolol combination induces a worse sexual function and a reduction of sex hormone,whereas felodipine-irbesartan combination does not impair sexual function and does not change hormone levels.
3. Oxidative stress decline after both combination regimens. Felodipine-irbesartan combination has a greater impact on oxidative stress indicators than felodipine-metoprolol combination.

DETAILED DESCRIPTION:
The effects of hypertension and its pharmacotherapy on sexual function are well known in men,although this topic remains unexplored in women.There is evidence suggests that some classes of antihypertensive drugs such as diuretics and beta-blockers have more negative impact on male sexual function than other classes such as calcium channel blockers(CCBs) and angiotensin-converting enzyme inhibitors(ACEI).Some data suggest that angiotensin Ⅱ antagonists（ARBs) not only do not exacerbate sexual function in males,but even improve it.

Treatment with multiple antihypertensive medications was often necessary to attain blood-pressure goals recommended by guidelines.More than two third of patients with 2 or 3 degree of essential hypertension require combination therapy at the beginning of treatment to avoid target organ damage and to minimize the accidence of adverse events.

CCBs were recommended by both JNC-7 and ESH / ESC 2007 hypertension guidelines as the basic for the treatment of hypertension.The purpose of this study is to compare the impacts of different CCB-based antihypertensive drugs combination on sexual behavior in both male and female patients with essential hypertension,thus provide evidences for physicians to increase patients adherence to the treatment regimens beside lowing blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential hypertension.
* Initial hypertension, or without taking any antihypertensive for at least one month.
* Sexual active.

Exclusion Criteria:

* Patients with secondary hypertension.
* Patients with malignant hypertension, coronary heart disease, diabetes, a history of syncope, bradycardia (heart rate <45 beats / min), atrioventricular block(Ⅱ or Ⅲ degree), sick sinus syndrome, congestive heart failure, a history of cerebral vascular accidents, serious hepatic and kidney dysfunction, a history of serious mental illness, pregnant, taking oral exogenous estrogens (including contraceptives), hysterectomy, breastfeeding, a history of alcohol or drug abuse, having serious conflict with sexual partner, severity sexual dysfunction.
* Patients refuse to answer questions, refuse to fill in the questionaires,or do not willing to take blood examination.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-10 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) | 48 weeks
  The Female Sexual Function Index (FSFI) is a multidimensional self-report scale for assessing sexual function in women.The FSFI hase been validated in women with various sexual disorders,and in non-dysfunctional controls showing good discriminant validity,internal consistency,and test-retest reliability.
International Index of Erectile Function(IIEF) | 48 weeks
  The 15-item International Index of Erectile Function (IIEF) was developed to diagnose the presence and severity of erectile dysfunction (ED).

SECONDARY OUTCOMES:
Change of Systolic Blood Pressure in 2 Weeks | 2 weeks
  The decrease of systolic blood pressure compared with baseline. Baseline is blood pressure in 0 week.
  BP is measured using a calibrated standard mercury sphygmomanometer.After the patient has been seated for 15 minutes,sitting BP is measured 2 times at 1- to 2-minutes intervals,The mean of 2 sitting BP measurements is used as the sitting BP value for that visit;If the difference between the 2 measurements is over 5mmHg,BP should be measured again, and the average of 3 measurements will be taken.
Change of Systolic Blood Pressure in 4 Weeks | 4 weeks
  The decrease of systolic blood pressure compared with baseline. Baseline is blood pressure in 0 week.
Change of Systolic Blood Pressure in 8 Weeks | 8 weeks
  The decrease of systolic blood pressure compared with baseline. Baseline is blood pressure in 0 week.
Change of Systolic Blood Pressure in 12 Weeks | 12 weeks
  The decrease of systolic blood pressure compared with baseline. Baseline is blood pressure in 0 week
Change of Systolic Blood Pressure in 24 Weeks | 24 weeks
  The decrease of systolic blood pressure compared with baseline. Baseline is blood pressure in 0 week.
Change of Systolic Blood Pressure in 48 Weeks | 48 weeks
  The decrease of systolic blood pressure compared with baseline. Baseline is blood pressure in 0 week
Change of Diastolic Blood Pressure in 2 Weeks | 2 weeks
  The decrease of diastolic blood pressure compared with baseline. Baseline is blood pressure in 0 week
Change of Diastolic Blood Pressure in 4 Weeks | 4 weeks
  The decrease of diastolic blood pressure compared with baseline. Baseline is blood pressure in 0 week
Change of Diastolic Blood Pressure in 8 Weeks | 8 weeks
  The decrease of diastolic blood pressure compared with baseline. Baseline is blood pressure in 0 week
Change of Diastolic Blood Pressure in 12 Weeks | 12 weeks
  The decrease of diastolic blood pressure compared with baseline. Baseline is blood pressure in 0 week.
Change of Diastolic Blood Pressure in 24 Weeks | 24 weeks
  The decrease of diastolic blood pressure compared with baseline. Baseline is blood pressure in 0 week.
Change of Diastolic Blood Pressure in 48 Weeks | 48 weeks
  The decrease of diastolic blood pressure compared with baseline. Baseline is blood pressure in 0 week.
Serum Estradiol in 24 Weeks | 24 weeks
  Fasting blood samples are taken at 8:00-10:00.After quiescence for 1h and centrifuged (3500rpm/min * 15min), serum samples are extracted and preserved in -80 ℃. Use hemiluminescent radioimmunoassay to detect the level of estradiol in serum sample.
Serum Estradiol in 48 Weeks | 48 weeks
Serum Testosterone in 24 Weeks | 24 weeks
  Fasting blood samples are taken at 8:00-10:00.After quiescence for 1h and centrifuged (3500rpm/min * 15min), serum samples are extracted and preserved in -80 ℃. Use hemiluminescent radioimmunoassay to detect the level of testosterone in serum sample.
Serum Testosterone in 48 Weeks | 48 weeks
Serum MDA in 24 Weeks | 24 weeks
  Among many oxidative stress biological indicators,malondialdehyde (MDA),the secondary products of lipid peroxidation,is the most representative and most studied polyunsaturated fatty acid peroxidation.
  Fasting blood samples are taken at 8:00-10:00.After quiescence for 1h and centrifuged (3500rpm/min * 15min), serum samples are extracted and preserved in -80 ℃. Use ELISA to detect the level of MDA in serum samples.
Serum MDA in 48 Weeks | 48 weeks
Serum 8-OHdG in 24 Weeks | 24 weeks
  Reactive oxygen species (ROS) produced either endogenously or exogenously can attack lipid, protein and nucleic acid simultaneously in the living cells. In nuclear and mitochondrial DNA, 8-hydroxydeoxyguanosine (8-OHdG) is produced during DNA repair and its measurement be useful as a marker of DNA lesion.
  Fasting blood samples are taken at 8:00-10:00.After quiescence for 1h and centrifuged (3500rpm/min * 15min), serum samples are extracted and preserved in -80 ℃. Use ELISA to detect the level of 8-OHdG in serum samples.
Serum 8-OHdG in 48 Weeks | 48 weeks
Serum HNE in 24 Weeks | 24 weeks
  4 - hydroxy-nonyl acid (HNE) is a strong toxicity end product of lipid peroxidation.
  Fasting blood samples are taken at 8:00-10:00.After quiescence for 1h and centrifuged (3500rpm/min * 15min), serum samples are extracted and preserved in -80 ℃. Use ELISA to detect the level of HNE in serum samples.
Serum HNE in 48 Weeks | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jing Yu, Professor, Study Chair — Lanzhou University Second Hospital
Locations (1):
- The Second Hospital of Lanzhou University, Lanzhou, Gansu, China

REFERENCES:
- [Background] WRITING GROUP MEMBERS; Lloyd-Jones D, Adams RJ, Brown TM, Carnethon M, Dai S, De Simone G, Ferguson TB, Ford E, Furie K, Gillespie C, Go A, Greenlund K, Haase N, Hailpern S, Ho PM, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott MM, Meigs J, Mozaffarian D, Mussolino M, Nichol G, Roger VL, Rosamond W, Sacco R, Sorlie P, Roger VL, Thom T, Wasserthiel-Smoller S, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation. 2010 Feb 23;121(7):e46-e215. doi: 10.1161/CIRCULATIONAHA.109.192667. Epub 2009 Dec 17. No abstract available. PMID 20019324
- [Background] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Background] Barzilay JI, Davis BR, Cutler JA, Pressel SL, Whelton PK, Basile J, Margolis KL, Ong ST, Sadler LS, Summerson J; ALLHAT Collaborative Research Group. Fasting glucose levels and incident diabetes mellitus in older nondiabetic adults randomized to receive 3 different classes of antihypertensive treatment: a report from the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). Arch Intern Med. 2006 Nov 13;166(20):2191-201. doi: 10.1001/archinte.166.20.2191. PMID 17101936
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Jamerson K, Weber MA, Bakris GL, Dahlof B, Pitt B, Shi V, Hester A, Gupte J, Gatlin M, Velazquez EJ; ACCOMPLISH Trial Investigators. Benazepril plus amlodipine or hydrochlorothiazide for hypertension in high-risk patients. N Engl J Med. 2008 Dec 4;359(23):2417-28. doi: 10.1056/NEJMoa0806182. PMID 19052124
- [Background] Dusing R. Effect of the angiotensin II antagonist valsartan on sexual function in hypertensive men. Blood Press Suppl. 2003 Dec;2:29-34. doi: 10.1080/08038020310021967. PMID 14761074
- [Background] Adverse reactions to bendrofluazide and propranolol for the treatment of mild hypertension. Report of Medical Research Council Working Party on Mild to Moderate Hypertension. Lancet. 1981 Sep 12;2(8246):539-43. PMID 6115999
- [Background] Grimm RH Jr, Grandits GA, Prineas RJ, McDonald RH, Lewis CE, Flack JM, Yunis C, Svendsen K, Liebson PR, Elmer PJ. Long-term effects on sexual function of five antihypertensive drugs and nutritional hygienic treatment in hypertensive men and women. Treatment of Mild Hypertension Study (TOMHS). Hypertension. 1997 Jan;29(1 Pt 1):8-14. doi: 10.1161/01.hyp.29.1.8. PMID 9039073
- [Background] Fogari R, Preti P, Derosa G, Marasi G, Zoppi A, Rinaldi A, Mugellini A. Effect of antihypertensive treatment with valsartan or atenolol on sexual activity and plasma testosterone in hypertensive men. Eur J Clin Pharmacol. 2002 Jun;58(3):177-80. doi: 10.1007/s00228-002-0456-3. Epub 2002 May 1. PMID 12107602
- [Background] Fogari R, Zoppi A, Corradi L, Mugellini A, Poletti L, Lusardi P. Sexual function in hypertensive males treated with lisinopril or atenolol: a cross-over study. Am J Hypertens. 1998 Oct;11(10):1244-7. doi: 10.1016/s0895-7061(98)00139-3. PMID 9799042
- [Background] Dusing R. Sexual dysfunction in male patients with hypertension: influence of antihypertensive drugs. Drugs. 2005;65(6):773-86. doi: 10.2165/00003495-200565060-00005. PMID 15819590
- [Background] Wassertheil-Smoller S, Blaufox MD, Oberman A, Davis BR, Swencionis C, Knerr MO, Hawkins CM, Langford HG. Effect of antihypertensives on sexual function and quality of life: the TAIM Study. Ann Intern Med. 1991 Apr 15;114(8):613-20. doi: 10.7326/0003-4819-114-8-613. PMID 2003706
- [Background] Fogari R, Preti P, Zoppi A, Corradi L, Pasotti C, Rinaldi A, Mugellini A. Effect of valsartan and atenolol on sexual behavior in hypertensive postmenopausal women. Am J Hypertens. 2004 Jan;17(1):77-81. doi: 10.1016/j.amjhyper.2003.08.016. PMID 14700518
- [Background] Meston CM. Validation of the Female Sexual Function Index (FSFI) in women with female orgasmic disorder and in women with hypoactive sexual desire disorder. J Sex Marital Ther. 2003 Jan-Feb;29(1):39-46. doi: 10.1080/713847100. PMID 12519665
- [Background] Wiegel M, Meston C, Rosen R. The female sexual function index (FSFI): cross-validation and development of clinical cutoff scores. J Sex Marital Ther. 2005 Jan-Feb;31(1):1-20. doi: 10.1080/00926230590475206. PMID 15841702
- [Background] Krapf JM, Simon JA. The role of testosterone in the management of hypoactive sexual desire disorder in postmenopausal women. Maturitas. 2009 Jul 20;63(3):213-9. doi: 10.1016/j.maturitas.2009.04.008. Epub 2009 May 31. PMID 19487090
- [Background] Basson R, Wierman ME, van Lankveld J, Brotto L. Summary of the recommendations on sexual dysfunctions in women. J Sex Med. 2010 Jan;7(1 Pt 2):314-26. doi: 10.1111/j.1743-6109.2009.01617.x. PMID 20092441
- [Background] Basson R. Pharmacotherapy for women's sexual dysfunction. Expert Opin Pharmacother. 2009 Jul;10(10):1631-48. doi: 10.1517/14656560903004184. PMID 19527189
- [Background] Berry C, Brosnan MJ, Fennell J, Hamilton CA, Dominiczak AF. Oxidative stress and vascular damage in hypertension. Curr Opin Nephrol Hypertens. 2001 Mar;10(2):247-55. doi: 10.1097/00041552-200103000-00014. PMID 11224701
- [Background] Lacy F, Kailasam MT, O'Connor DT, Schmid-Schonbein GW, Parmer RJ. Plasma hydrogen peroxide production in human essential hypertension: role of heredity, gender, and ethnicity. Hypertension. 2000 Nov;36(5):878-84. doi: 10.1161/01.hyp.36.5.878. PMID 11082160
- [Background] Agarwal A, Gupta S, Sharma R. Oxidative stress and its implications in female infertility - a clinician's perspective. Reprod Biomed Online. 2005 Nov;11(5):641-50. doi: 10.1016/s1472-6483(10)61174-1. PMID 16409717
- [Background] Vlachopoulos C, Aznaouridis K, Ioakeimidis N, Rokkas K, Tsekoura D, Vasiliadou C, Stefanadi E, Askitis A, Stefanadis C. Arterial function and intima-media thickness in hypertensive patients with erectile dysfunction. J Hypertens. 2008 Sep;26(9):1829-36. doi: 10.1097/HJH.0b013e3283050886. PMID 18698219
- [Background] Dincer Y, Sekercioglu N, Pekpak M, Gunes KN, Akcay T. Assessment of DNA oxidation and antioxidant activity in hypertensive patients with chronic kidney disease. Ren Fail. 2008;30(10):1006-11. doi: 10.1080/08860220802422044. PMID 19016153
- [Background] Agarwal A, Gupta S, Sikka S. The role of free radicals and antioxidants in reproduction. Curr Opin Obstet Gynecol. 2006 Jun;18(3):325-32. doi: 10.1097/01.gco.0000193003.58158.4e. PMID 16735834
- [Background] Ono H, Minatoguchi S, Watanabe K, Yamada Y, Mizukusa T, Kawasaki H, Takahashi H, Uno T, Tsukamoto T, Hiei K, Fujiwara H. Candesartan decreases carotid intima-media thickness by enhancing nitric oxide and decreasing oxidative stress in patients with hypertension. Hypertens Res. 2008 Feb;31(2):271-9. doi: 10.1291/hypres.31.271. PMID 18360047
- [Background] de la Sierra A, Larrousse M. Endothelial dysfunction is associated with increased levels of biomarkers in essential hypertension. J Hum Hypertens. 2010 Jun;24(6):373-9. doi: 10.1038/jhh.2009.91. Epub 2009 Nov 26. PMID 19960026
- [Background] Rothwell PM, Howard SC, Dolan E, O'Brien E, Dobson JE, Dahlof B, Poulter NR, Sever PS; ASCOT-BPLA and MRC Trial Investigators. Effects of beta blockers and calcium-channel blockers on within-individual variability in blood pressure and risk of stroke. Lancet Neurol. 2010 May;9(5):469-80. doi: 10.1016/S1474-4422(10)70066-1. Epub 2010 Mar 11. PMID 20227347
- [Derived] Ma R, Yu J, Xu D, Yang L, Lin X, Zhao F, Bai F. Effect of felodipine with irbesartan or metoprolol on sexual function and oxidative stress in women with essential hypertension. J Hypertens. 2012 Jan;30(1):210-6. doi: 10.1097/HJH.0b013e32834e1e2e. PMID 22134388